CLINICAL TRIAL: NCT02506790
Title: Phase II Multicenter Randomized Study to Compare Neoadjuvant Toremifene With Melatonin or Metformin Versus Toremifene in the Therapy of Locally Advanced Breast
Brief Title: Neoadjuvant Toremifene With Melatonin or Metformin in Locally Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBC 2
Record Dates: First submitted 2015-07-17; First posted 2015-07-23 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Melatonin, metformin, toremifene
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Melatonin; Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Toremifene and metformin (Experimental): Toremifene 60 mg daily with metformin 850 mg BID
  Interventions: Drug: metformin; Drug: Toremifene
- Toremifene and melatonin (Experimental): Toremifene 60 mg daily with melatonin 3 mg before sleep daily
  Interventions: Drug: Melatonin; Drug: Toremifene
- Toremifene (Active Comparator): Toremifene 60 mg daily
  Interventions: Drug: Toremifene

INTERVENTIONS:
Drug: metformin
  Other Names: siofor 850
  Arms: Toremifene and metformin
Drug: Melatonin
  Other Names: melaxen
  Arms: Toremifene and melatonin
Drug: Toremifene
  Other Names: farestone

SUMMARY:
This study evaluates the addition melatonin and metformin to toremifene in the treatment of locally advanced breast cancer. Third of patients will receive toremifene, other third will receive combination of melatonin and toremifene and other patients will receive combination of metformin and toremifene.

DETAILED DESCRIPTION:
The management of locally advanced breast cancer is complicated issue. Neoadjuvant treatment is often needed to downstage locally advanced ER positive BC tumors prior to surgery. However, many patients do not achieved objective response on treatment. The ability of melatonin and metformin to decrease side effects of chemotherapy had been investigated, moreover, several studies confirm, that this drugs in combination with conventional anti - estrogen treatment may increase objective response. But, this data is still controversial. We hypothesizes that the combinations of melatonin and metformin with conventional anti - estrogen such as toremifene could be more effective than toremifene alone in terms of response rate.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18.
* Obtained Inform Concent.
* Morphologically confirmed breast cancer stage IIB, IIIA, IIIB, IIIC ER positive.
* Eastern Collaborative Oncology Group Performance Status Scale 0-2.
* Expected survival > 6 month.
* Adequate liver and bone marrow function.

Exclusion Criteria:

* Systemic treatment for breast cancer.
* Stage IV disease.
* Evidence of liver and bone marrow clinically meaningful disfunction.
* Severe uncontrolled concomitant conditions and diseases.
* Pregnancy or lactation.
* Second malignancy.
* Diabetes mellitus requiring drug therapy.
* Any condition preventing study participation by investigators opinion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Response rate | 4 months after FPFV
  Response will evaluate by RECIST criteria
Pathomorphological response | 4 months after FPFV
  Pathomorphological response will assess after surgery by Miller and Payne Scale

SECONDARY OUTCOMES:
Adverse events incidence | Until 30 days after last patient treatment visit
  Incidence of AE classified using NCI Common Terminology Criteria for AE v4

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir F Semiglazov, MD,PhD, DSc, Professor, Study Director — N.N. Petrov Research Institute Of Oncology; Tatiana Y Semiglazova, MD, PhD, DSc, Principal Investigator — N.N. Petrov Research Institute Of Oncology
Locations (1):
- N.N. Petrov Research Institute of Oncology Clinical Diagnostic Department, Saint Petersburg, Russia